CLINICAL TRIAL: NCT06238128
Title: Developing and Testing the Opioid Rapid Response System
Brief Title: Opioid Rapid Response System: Naloxone Training in Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Hye Jeong Choi, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2097714
Record Dates: First submitted 2023-08-21; First posted 2024-02-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Opioid Overdose
Keywords: naloxone training; Community-engagement
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORRS training group (Experimental): Online Naloxone training
  Interventions: Behavioral: Opioid Rapid Resonse System (ORRS) training
- Waitlist group (Sham Comparator): Participants will receive non-active opioid overdose response training. Investigators will provide online training about opioid prevalence in US, opioid mechanism, side effect, and addiction. However, Investigators do not provide any knowledge about opioid overdose management and naloxone in this training.
  Once the project is completed, participants will receive online Naloxone training.
  Interventions: Behavioral: Non-active opioid overdose response training

INTERVENTIONS:
Behavioral: Opioid Rapid Resonse System (ORRS) training — ORRS is on online system to train citizen responders to administer NARCAN to save the lives of opioid overdose victims. It capitalizes on the innovative PulsePoint technology to connect responders to overdose events. PulsePoint is an app that connects 911 requesting assistance for cardiac arrests to responders with Cardiopulmonary Resuscitation (CPR) training. ORRS allows us to partner with PulsePoint users to expand its reach to opioid overdoses, which share the need for a quick response that emergency responders are often unable to provide. ORRS has the advantage of expanding the population of responders with NARCAN, rescue breathing, and CPR training that can be connected to overdose events, increasing the likelihood of saving overdose victims' lives through a quick, efficient response. ORRS is delivered through an interactive, digital platform containing sequential, multi-media modules.
  Arms: ORRS training group
Behavioral: Non-active opioid overdose response training — Investigators will provide online training about opioid prevalence in US, opioid mechanism, side effect, and addiction. However, Investigators do not provide any knowledge about opioid overdose management and naloxone in this training.
  Once the project is completed, participants will receive online Naloxone training.
  Arms: Waitlist group

SUMMARY:
The pervasive impact of the opioid epidemic has touched all layers of society for the past two decades, resulting in over 115 deaths daily and imposing annual costs of $78.5 billion. Responding swiftly to overdoses, akin to various medical emergencies, poses a significant challenge, particularly in geographically dispersed rural areas and densely populated urban settings. Effectively delivering the life-saving drug naloxone, which counteracts the effects of overdoses, necessitates a well-coordinated and cost-efficient response system.

Simply opting for widespread distribution of naloxone, even with citizen involvement, proves to be a financially burdensome approach when compared to more targeted strategies. Moreover, obstacles such as limited access, inadequate or unavailable naloxone training, and delayed response times from emergency responders compound the problem. Addressing these issues, the proposed Opioid Rapid Response System (ORRS) project seeks to advance prevention science by adopting an innovative approach that incorporates technology and contemporary communication theory.

The primary objective of the ORRS project is to mitigate opioid overdose deaths by enlisting and training citizens to administer naloxone in response to such events. Leveraging the PulsePoint health app, which connects citizens to cardiac events, the ORRS project will extend its capabilities to respond to overdose incidents. This initiative involves comprehensive development of ORRS, followed by a randomized clinical trial on a national scale to assess its effectiveness. The study aims to contribute to both prevention and implementation science by identifying optimal recruitment strategies and testing a model of online training. In pursuit of these objectives, the study is guided by the following Specific Aims:

SA 1: Refine and complete the development of ORRS. SA 2: Conduct a randomized clinical trial to evaluate the effectiveness of the intervention. SA 3: Prepare ORRS for dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Citizens who live in participating PulsePoint communities
* Must to be 18 and older
* Must be fluent in English
* Must have access to the mobile data and able to download and use apps in a smartphone

Exclusion Criteria:

* Citizens who do not live in participating PulsePoint communities
* Under 18-year-old
* Citizens who are not fluent in English
* Citizens who do not have access to mobile data and unable to download and use apps in a smartphone.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Knowledge of overdose sign | up to 2 weeks
  Investigators will use a subset of Opioid Overdose Knowledge Scale (OOKS) to measure through a forced choice scale with each choice coded as correct (=1) or incorrect (=0). Higher score indicated greater knowledge of overdose sign.
Knowledge of overdose management | up to 2 weeks
  Investigators will use a subset of Opioid Overdose Knowledge Scale (OOKS) to measure through a forced choice scale with each choice coded as correct (=1) or incorrect (=0). Higher score indicated greater knowledge of overdose management.
Self-Efficacy toward intervening opioid overdose | up to 2 weeks
  Investigators will modify self-efficacy scale developed and theorized by Bandura (2005). Response options are from 0 (no confident) to 100 (highly confident). Higher score indicates greater self-efficacy
Response efficacy about intervening opioid overdose | up to 2 weeks
  Investigators will develop and measure how participants perceive the effectiveness of activities to intervene opioid overdose events in communities. Response options are from 0 (not effective) to 100 (highly effective). Higher score indicate greater response efficacy.
Concerns related to overdose management | up to 2 weeks
  Investigators will use a subset of Opioid Overdose Attitude Scale (OOAS) with 5 point scale (1: strongly disagree ~5: strongly agree). Higher score indicates the greater concerns.
Intent to intervene opioid overdose events in communities | up to 2 weeks
  Investigators will use behavioral intention scale developed by in the opioid training literature (Hecht et al., 2023) to measure intent to intervene opioid overdose events in communities (e.g., administering Narcan). Response options are from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicates grater intention to intervene opioid overdose events in communities.
The number of days per week, on average, to carry Narcan | Up to 6 months
  Single item: how many days per week, on average, participants carry Narcn
Number of Participants to response to overdose events from PulsePoint app. | Up to 6 months
  Single item: whether participant response to overdose events from PulsePoint notifications/alerts
Number of participants to administer Narcan | Up to 6 months
  Single item: Whether participant administer Narcan to respond opioid overdose events in communities.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jeong Choi, Principal Investigator — Univeristy of Missouri; Michael Hecht, Principal Investigator — Real Prevention
Locations (1):
- Ewald & Wasserman Research Consultants, LLC, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Because this study is funded as a part of NIH HEAL initiative, investigators will follow the HEAL data sharing policy.
Supporting Information: Study Protocol, ICF
Time Frame: When project is completed.

REFERENCES:
- [Derived] Carr DL, Hecht ML, Shiota MN, Zalake M, Krieger J, Choi HJ. Protocol for a national randomized controlled trial evaluating the Opioid Rapid Response System for overdose death prevention. Contemp Clin Trials. 2025 Mar;150:107835. doi: 10.1016/j.cct.2025.107835. Epub 2025 Feb 3. PMID 39909302